CLINICAL TRIAL: NCT01199809
Title: A Multi-center, Randomized, Observer-blinded, Multiple-Ascending-Dose, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO5310074 Following Multiple Intravenous Administrations in Subjects With Psoriatic Arthritis
Brief Title: A Study of RO5310074 in Patients With Psoriatic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP22713; 2011-001133-16 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO5310074
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — multiple doses
  Arms: 2
Drug: RO5310074 — multiple ascending doses
  Arms: 1

SUMMARY:
This randomized, double-blind. placebo-controlled study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of RO5310074 in patients with psoriatic arthritis who have or have had an inadequate response to oral disease-modifying antirheumatic drugs (DMARDs) or non-steroidal anti-rheumatic drugs (NSAIDs). Patients will be randomized in cohorts to receive either 6 intravenous doses of RO5310074 or placebo. Anticipated time on study treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 - 75 years of age
* Diagnosis of Psoriatic Arthritis (Moll and Wright or CASPAR criteria) of >/= 6 months duration
* Have >/= 3 swollen and >/= 3 tender joints
* Inadequate response to a current or previous oral DMARD or NSAID therapy
* Current oral DMARDs must be at stable dose for the appropriate duration (e.g. 14 days for sulfasalazine and 28 days for methotrexate or oral steroids)
* NSAIDs up to maximum recommended dose are permitted if at stable dose for at least 14 days prior to first dose of study drug, but not more than one NSAID simultaneously (except for low-dose aspirin for cardioprotection)
* Body mass index (BMI) 18 - 42 kg/m2 inclusive

Exclusion Criteria:

* Previous prolonged treatment with a biologic DMARD; use of biologic DMARD within 3 months or 5 times its elimination half-live (whichever is longer) prior to first dose of study drug
* Previous use of B-cell depleting biologic DMARDs
* Any previous treatment with alkylating agents such a cyclophosphamide or chlorambucil or with total lymphoid irradiation
* History of or current inflammatory joint disease other than psoriatic arthritis; Gout or pseudogout that is current or has been active within the past 6 months
* Positive for hepatitis B, hepatitis C or HIV infection
* Any acquired or congenital immune deficiency or history of disease known to cause significant alteration in immunologic function
* Acute clinically significant infection in the 6 weeks prior to administration of study drug, history or presence of chronic infection, or history of recurrent infection as an adult

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 25 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax, t1/2, AUC, Vss, CL) | 12 weeks
Pharmacodynamics (anti-drug-antibodies) | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (6):
  - Anniston, Alabama
  - Los Angeles, California
  - Miami, Florida
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
- Australia (2):
  - Melbourne, Victoria
  - Nedlands, Western Australia
- Christchurch, New Zealand